CLINICAL TRIAL: NCT02152631
Title: JUNIPER: A Randomized Phase 3 Study of Abemaciclib Plus Best Supportive Care Versus Erlotinib Plus Best Supportive Care in Patients With Stage IV NSCLC With a Detectable KRAS Mutation Who Have Progressed After Platinum-Based Chemotherapy
Brief Title: A Study of Abemaciclib (LY2835219) in Participants With Previously Treated KRAS Mutated Lung Cancer
Acronym: JUNIPER
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15296; I3Y-MC-JPBK (Other: Eli Lilly and Company); 2013-004662-33 (EudraCT Number)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2014-05-23; First posted 2014-06-02 (Estimated); Results first posted 2018-12-12 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Therapy, Platinum, Kras +
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — abemaciclib; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abemaciclib (Experimental): 200 milligrams (mg) abemaciclib administered, orally, every 12 hours plus best supportive care (BSC) on Days 1 to 28 (28 day cycles).
  Interventions: Drug: Abemaciclib
- Erlotinib (Active Comparator): 150 mg erlotinib administered, orally, every 24 hours plus BSC on Days 1 to 28 (28 day cycles).
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219
  Arms: Abemaciclib
Drug: Erlotinib — Administered orally
  Arms: Erlotinib

SUMMARY:
The main purpose of this study is to evaluate how safe and effective the study drug known as abemaciclib is in participants with lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have confirmed diagnosis of stage IV non-small cell lung cancer (NSCLC) according to the American Joint Committee on Cancer Staging Handbook.
* Determined to have detectable mutations in codons 12 or 13 of the kirsten rat sarcoma (KRAS) oncogene by an investigational assay at the study central laboratory. A KRAS positive mutation result in codons 12 or 13 of the KRAS oncogene from tumor tissue per local laboratory will be permitted in no more than 10% of randomized participants.
* Have progressed after platinum-based chemotherapy (with or without maintenance therapy) AND have received one additional therapy which may include an immune checkpoint inhibitor or other anti-cancer therapy for advanced and/or metastatic disease OR is judged by the physician as ineligible for further standard second-line chemotherapy. Participants who have progressed after platinum-based chemotherapy and an immune checkpoint inhibitor (immunotherapy) e.g. pembrolizumab or nivolumab alone or in combination with other agents are eligible.
* Have measureable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
* Have a performance status (PS) of 0 to 1 on the Eastern Cooperative Oncology Group (ECOG) scale.
* Have discontinued all previous therapies for cancer (including chemotherapy, radiotherapy, immunotherapy, and investigational therapy) for at least 21 days for myelosuppressive agents or 14 days for nonmyelosuppressive agents prior to receiving study drug.

Exclusion Criteria:

* Have received treatment with a drug that has not received regulatory approval for any indication within 14 or 21 days of the initial dose of study drug for a nonmyelosuppressive or myelosuppressive agent, respectively.
* Have a personal history of any of the following conditions: presyncope or syncope of either unexplained or cardiovascular etiology, ventricular arrhythmia (including but not limited to ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
* Have the presence of unstable central nervous system (CNS) metastasis. History of CNS metastasis or stable CNS metastases is allowed (no longer requiring active therapy such as steroid medications). Participants with a history of CNS metastases must have a brain scan (for example, magnetic resonance imaging [MRI]) within 28 days of randomization to document stability, even if there have been no changes in symptoms.
* Have previously completed or withdrawn from this study or any other study investigating a cyclin-dependent kinase 4 (CDK4) and cyclin-dependent kinase 6 (CDK6) inhibitors, or have received treatment with a prior CDK4 and CDK6 inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2014-10-03 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (209):
- United States (54):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - St. Bernards Medical Center, Jonesboro, Arkansas
  - City of Hope National Medical Center, Duarte, California
  - University of California - San Diego, La Jolla, California
  - Loma Linda University School of Medicine, Loma Linda, California
  - CBCC Global Research, Inc., Los Angeles, California
  - Central Coast Medical Oncology Corporation, Los Angeles, California
  - Fort Wayne Oncology & Hematology, Los Angeles, California
  - SMO TRIO -Translational Research, Los Angeles, California
  - St. Joseph Heritage Medical Group, Los Angeles, California
  - UCLA Department of Medicine-Hematology/Oncology, Los Angeles, California
  - Cancer Care Associates Medical Group, Los Angeles, California
  - Dignity Health Care Institute, Sacramento, California
  - Alegent Immanuel Cancer Center, Englewood, Colorado
  - Jewish Hospital, Englewood, Colorado
  - Oncology Hematology West, Englewood, Colorado
  - SMO Catholic Health Initiatives, Englewood, Colorado
  - St Joseph Cancer Center, Englewood, Colorado
  - St. Francis Medical Center, Englewood, Colorado
  - Medical Oncology Hematology Consultants, Newark, Delaware
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Halifax Medical Center, Daytona Beach, Florida
  - Memorial Cancer Institute, Pembroke Pines, Florida
  - H Lee Moffitt Cancer Center, Tampa, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Cancer Center of Kansas, P.A., Wichita, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Metro-West and Greater Boston CNS Research, Framingham, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mercy Medical Research Institute, Springfield, Missouri
  - Billings Clinic Research Center, Billings, Montana
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Broome Oncology, Johnson City, New York
  - Weill Cornell Medical College, New York, New York
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Oklahoma Cancer Specialists & Research Institute, LLC, Tulsa, Oklahoma
  - Providence Cancer Center Oncology Hematology Care, Portland, Oregon
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Roper St. Francis Healthcare, Charleston, South Carolina
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Chattanooga Oncology Hematology Associates, Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - Virginia Commonwealth University, Richmond, Virginia
  - Kadlec Clinical Hematology & Oncology, Kennewick, Washington
  - Swedish Medical Center, Seattle, Washington
  - Cancer Care Northwest, Valley, Washington
- Argentina (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Berazategui
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ciudad Autonoma Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rosario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Rosario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Viedma
- Austria (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Graz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Linz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Linz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salzburg
- Brazil (8):
  - Associação Hospital de Caridade Ijuí, Ijuí
  - Hospital Bruno Born, Lajeados
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto Alegre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio de Janeiro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salvador
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sao Jose Rio Preto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, São Paulo
  - Fundação Antonio Prudente - Hospital do Câncer A.C Camargo, São Paulo
- Canada (6):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Calgary
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Edmonton
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Montreal
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Toronto
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Vancouver
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Winnipeg
- China (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changchun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chengdu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haikou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hefei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanning
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shenyang
- France (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bron
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Dijon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grenoble
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poitiers
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rennes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Saint-Brieuc
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Priest-en-Jarez
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vantoux
- Germany (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gera
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Großhansdorf
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Immenhausen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nuremberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Regensburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rosenheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tübingen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulm
- Greece (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heraklion
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pátrai
- Israel (6):
  - Soroka Medical Center, Beersheba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Holon
  - Hadassah Medical Center - Ein Karem, Jerusalem
  - Meir Medical Center, Kfar Saba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Petah Tikva
  - Sheba Medical Center, Tel Litwinsky
- Italy (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Catania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Livorno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
- Japan (32):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amagasaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Asahikawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bunkyō City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Habikino
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hirakata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hiroshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanazawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kashiwa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kishiwada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kitaadachi-Gun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kobe
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kōtoku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kurashiki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Matsuyama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagasaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagoya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Natori
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sakai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sendai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shinjuku-ku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sunto-Gun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ube
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Utsunomiya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wakayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yokohama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yonago
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yufu-shi
- Poland (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olsztyn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Radom
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szczecin
- VA Caribbean Healthcare System, San Juan, Puerto Rico
- Romania (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baia Mare
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Craiova
- Russia (9):
  - Arkhangelsk Regional Clinical Oncology Dispensary, Arkhangelsk
  - Private clinic "Evimed", Chelyabinsk
  - Krasnodar regional clinical hospital # 1 n. a. S. V. Ochapovskogo, Krasnodar
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kursk
  - Russian oncological scientific centre n.a. N.N. Blokhin of RAMS, Moscow
  - St-Petersburg scientifical practical center of specialized kinds of medical care (oncological), Saint Petersburg
  - Saint-Petersburg city clinical oncology dispensary, Saint Petersburg
  - Republic clinical oncology dispensary of MoH of Bashkortostan Republic, Ufa
  - Volgograd regional clinical oncology dispensary, Volzhskiy
- South Korea (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goyang-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Incheon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seowon-Gu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suwon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulsan
- Spain (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., A Coruña
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., L'Hospitalet de Llobregat
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Málaga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
- Taiwan (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiayi City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaohsiung City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tainan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zhonghe
- Turkey (Türkiye) (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ankara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Antalya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edirne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Istanbul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Izmir
- Ukraine (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dnipropetrovsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kharkiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kryvyi Rih
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lutsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poltava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sumy
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Uzhhorod
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vinnitsa

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Goldman JW, Mazieres J, Barlesi F, Dragnev KH, Koczywas M, Goskel T, Cortot AB, Girard N, Wesseler C, Bischoff H, Nadal E, Park K, Lu S, Taus A, Cobo M, Estrem ST, Wijayawardana SR, Turner K, Oakley GJ 3rd, Hurt KC, Chiang AY, Hossain AM, John WJ, Paz-Ares L. A Randomized Phase III Study of Abemaciclib Versus Erlotinib in Patients with Stage IV Non-small Cell Lung Cancer With a Detectable KRAS Mutation Who Failed Prior Platinum-Based Therapy: JUNIPER. Front Oncol. 2020 Oct 26;10:578756. doi: 10.3389/fonc.2020.578756. eCollection 2020. PMID 33194700
- [Derived] Goldman JW, Shi P, Reck M, Paz-Ares L, Koustenis A, Hurt KC. Treatment Rationale and Study Design for the JUNIPER Study: A Randomized Phase III Study of Abemaciclib With Best Supportive Care Versus Erlotinib With Best Supportive Care in Patients With Stage IV Non-Small-Cell Lung Cancer With a Detectable KRAS Mutation Whose Disease Has Progressed After Platinum-Based Chemotherapy. Clin Lung Cancer. 2016 Jan;17(1):80-4. doi: 10.1016/j.cllc.2015.08.003. Epub 2015 Aug 18. PMID 26432508
- See also: A Study of Abemaciclib (LY2835219) in Participants With Previously Treated KRAS Mutated Lung Cancer — https://trials.lillytrialguide.com/en-US/trial/6apfdhnUhG22E8AcMmSCCC

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers are defined as those participants who had progressive disease, death due to any cause or alive and on study at the end of study, but off treatment.
Period: Overall Study
Arm/Group | Abemaciclib | Erlotinib
Started | 270 | 183
Received at Least One Dose of Study Drug | 265 | 175
Off Treatment | 246 | 172
Death Due to Any Cause | 30 | 20
Progressive Disease | 174 | 137
Completed | 204 | 157
Not Completed | 66 | 26
Not completed — Adverse Event | 32 | 4
Not completed — Withdrawal by Subject | 13 | 16
Not completed — Noncompliance with study drug | 1 | 0
Not completed — Physician Decision | 1 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — On Treatment | 19 | 3

BASELINE CHARACTERISTICS:
Groups:
- Abemaciclib: 200 mg abemaciclib administered, orally, every 12 hours plus BSC on Days 1 to 28 (28 day cycles).
- Total: Total of all reporting groups
Arm/Group | Abemaciclib | Erlotinib | Total
Number analyzed (Participants) | 270 | 183 | 453
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (8.9) | 62.9 (8.4) | 62.5 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 74 | 181
  Male | 163 | 109 | 272
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 12 | 25
  Not Hispanic or Latino | 197 | 132 | 329
  Unknown or Not Reported | 60 | 39 | 99
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 56 | 41 | 97
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 165 | 106 | 271
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 45 | 32 | 77
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 1 | 2 | 3
  Romania | 7 | 7 | 14
  United States | 44 | 30 | 74
  Japan | 22 | 17 | 39
  Ukraine | 6 | 5 | 11
  Russia | 8 | 4 | 12
  Spain | 26 | 13 | 39
  Greece | 1 | 6 | 7
  Canada | 4 | 4 | 8
  Austria | 0 | 2 | 2
  South Korea | 13 | 13 | 26
  Turkey | 21 | 8 | 29
  China | 7 | 4 | 11
  Taiwan | 12 | 7 | 19
  Brazil | 7 | 5 | 12
  Poland | 6 | 2 | 8
  Italy | 5 | 12 | 17
  Israel | 5 | 1 | 6
  France | 35 | 32 | 67
  Germany | 30 | 14 | 44

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS defined as from randomization date to the date of death due to any cause. For each participant who is not known to have died as of the data-inclusion cutoff date for overall survival analysis, OS time was censored on the last date the participant is known to be alive.
Time Frame: From Randomization Date to Date of Death from Any Cause (Up to 32 Months)
Population: All randomized participants. 81 participants were censored in the Abemaciclib arm and 56 participants were censored in the Erlotinib arm.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abemaciclib | Erlotinib
Number analyzed (Participants) | 270 | 183
months | 7.4 [6.5 to 8.8] | 7.8 [6.4 to 9.5]
Statistical Analysis 1: Comparison: Abemaciclib vs Erlotinib; The stratification factors used in the analysis were: number of prior chemotherapy regimens (1 versus 2), Eastern Cooperative Oncology Group (ECOG) Performance Score (PS) (0 versus 1), gender (male versus female), and kirsten rat sarcoma (KRAS) mutation (GLY12CYS [G12C] vs. all others); Test type: Superiority; p = 0.771, Stratified Log-Rank; Hazard Ratio (HR) = 0.968, 95% CI 2-sided [0.768 to 1.219] — Hazard Ratio (HR) was estimated based on Stratified Cox proportional hazard model

2. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) (Objective Response Rate [ORR])
Description: ORR was the percentage of participants achieving a best overall response (BOR) of complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions.
Time Frame: From Randomization Date to Objective Progression (Up to 32 Months)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abemaciclib | Erlotinib
Number analyzed (Participants) | 270 | 183
percentage of participants | 8.9 [5.5 to 12.3] | 2.7 [0.4 to 5.1]
Statistical Analysis 1: Comparison: Abemaciclib vs Erlotinib; Stratified by number of prior chemotherapy regimens (1 versus 2), ECOG PS (0 versus 1), gender (male versus female), and KRAS mutation (GLY12CYS [G12C] vs. all others); Test type: Superiority; p = 0.010, Cochran-Mantel-Haenszel

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS defined as the from randomization date to the first evidence of disease progression as defined by RECIST v1.1 or death from any cause. Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. If a participant does not have a complete baseline disease assessment, then the PFS time was censored at the date of first dose, regardless of whether or not objectively determined disease progression or death has been observed for the participant. If a participant was not known to have died or have objective progression as of the data inclusion cutoff date for the analysis, the PFS time was censored at the last adequate tumor assessment date.
Time Frame: From Randomization Date until Disease Progression or Death from Any Cause (Up to 32 Months)
Population: All randomized participants. 36 participants were censored in the abemaciclib arm and 24 were censored in the erlotinib arm.
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Abemaciclib | Erlotinib
Number analyzed (Participants) | 270 | 183
months | 3.6 [2.8 to 3.8] | 1.9 [1.9 to 2.0]
Statistical Analysis 1: Comparison: Abemaciclib vs Erlotinib; Test type: Superiority; p < 0.000001, Stratified Log-Rank; Hazard Ratio (HR) = 0.583, 95% CI 2-sided [0.470 to 0.723]

4. Secondary Outcome: Change From Baseline in MD Anderson Symptom Inventory-Lung Cancer (MDASI-LC) Score
Description: The MDASI-LC included 22 items + 3 additional trial-specific items, resulting in 6 collected and reported single-construct scores including core symptoms (13-item), interference (6-item), lung cancer (3-item), and trial-specific single outcomes for headache, diarrhea, and rash. A 2-construct composite core + lung cancer symptom (16-item) score was calculated. Data for all 7 scores were collected by an 11-point numeric rating scale anchored at 0 (not present or does not interfere) and 10 (as bad as you can imagine or interfered completely). The measurement range was 10 (maximum score-minimum score). Mixed Model Repeated Measure (MMRM) regression with covariates for treatment, visit, treatment*visit, and baseline score predicted between-group Least Squares (LS) mean differences from baseline. Group-level negative change from baseline indicated group improvement.
Time Frame: From Randomization Date through End of Study (Up to 32 Months)
Population: All randomized participants for cycles which at least 25% of participants in each arm have a score. MDASI-LC population included all randomized participants who completed at least 1 baseline assessment followed by at least 1 MDASI-LC result.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Abemaciclib | Erlotinib
Number analyzed (Participants) | 270 | 183
units on a scale
  Headache | 0.20 (0.11) | 0.27 (0.15)
  Diarrhea | 1.91 (0.17) | 1.32 (0.23)
  Rash | 0.65 (0.17) | 3.05 (0.22)
  Mean Core Symptom Severity | 0.49 (0.10) | 0.73 (0.13)
  Mean Interference | 0.70 (0.14) | 0.85 (0.18)
  Mean Lung Cancer Symptom Severity | 0.16 (0.09) | 0.23 (0.12)
  Mean Core Plus Lung Cancer Symptom Severity | 0.44 (0.09) | 0.65 (0.12)
Statistical Analysis 1: Comparison: Abemaciclib vs Erlotinib; Headache; Test type: Superiority; p = 0.698, Mixed Models Analysis; Analyzed by Type 3 sums of squares, model covariates included Treatment + Visit + Treatment*Visit + Baseline; LS Mean Change Difference = -0.07, 95% CI 2-sided [-0.44 to 0.29], Standard Error of Mean 0.19
Statistical Analysis 2: Comparison: Abemaciclib vs Erlotinib; Diarrhea; Test type: Superiority; p = 0.038, Mixed Models Analysis; Analyzed by Type 3 sums of squares, model covariates included Treatment + Visit + Treatment*Visit + Baseline; LS Mean Change Difference = 0.59, 95% CI 2-sided [0.03 to 1.15], Standard Error of Mean 0.28
Statistical Analysis 3: Comparison: Abemaciclib vs Erlotinib; Rash; Test type: Superiority; p < .001, Mixed Models Analysis; Analyzed by Type 3 sums of squares, model covariates included Treatment + Visit + Treatment*Visit + Baseline; LS Mean Change Difference = -2.40, 95% CI 2-sided [-2.94 to -1.86], Standard Error of Mean 0.27
Statistical Analysis 4: Comparison: Abemaciclib vs Erlotinib; Mean Core Symptom Severity; Test type: Superiority; p = 0.142, Mixed Models Analysis; Analyzed by Type 3 sums of squares, model covariates included Treatment + Visit + Treatment*Visit + Baseline; LS Mean Change Difference = -0.24, 95% CI 2-sided [-0.56 to 0.08], Standard Error of Mean 0.16
Statistical Analysis 5: Comparison: Abemaciclib vs Erlotinib; Mean Interference; Test type: Superiority; p = 0.514, Mixed Models Analysis; Analyzed by Type 3 sums of square, model covariates included Treatment + Visit + Treatment*Visit + Baseline; LS Mean Change Difference = -0.15, 95% CI 2-sided [-0.59 to 0.30], Standard Error of Mean 0.23
Statistical Analysis 6: Comparison: Abemaciclib vs Erlotinib; Mean Lung Cancer; Test type: Superiority; p = 0.646, Mixed Models Analysis; Analyzed by Type 3 sums of squares, model covariates included Treatment + Visit + Treatment*Visit + Baseline; LS Mean Change Difference = -0.07, 95% CI 2-sided [-0.37 to 0.23], Standard Error of Mean 0.15
Statistical Analysis 7: Comparison: Abemaciclib vs Erlotinib; Mean Core Plus Lung Cancer; Test type: Superiority; p = 0.188, Mixed Models Analysis; Analyzed by Type 3 sums of squares, model covariates included Treatment + Visit + Treatment*Visit + Baseline; LS Mean Change Difference = -0.20, 95% CI 2-sided [-0.51 to 0.10], Standard Error of Mean 0.15

5. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve During 1 Dosing Interval at Steady State
Description: PK is determined by the area under the plasma concentration versus time curve during 1 dosing interval at steady state
Time Frame: Day 1 of Cycle 1 through Cycle 3 (28 Day Cycles)
Population: All randomized participants who received Abemaciclib and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram/milliliter (h*ng/mL)
Arm/Group | Abemaciclib
Number analyzed (Participants) | 265
Hour*nanogram/milliliter (h*ng/mL) | 3350 (52)

6. Secondary Outcome: Change From Baseline in European Quality of Life - 5 Dimensions - 5 Level (EQ-5D-5L) Score
Description: There are 5 response levels on a good-to-bad continuum of 1-5 corresponding to none, slight, moderate, severe, and extreme/unable to. The EuroQol-developed crosswalk method was used to convert the EQ-5D-5L,using United Kingdom (UK) weights, health dimensions(mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) into a single index value; the dimensions are not separately scored. The index is marked missing when ≥1 dimensions are missing. The index scores for the response patterns were anchored on full health to dead with negative values assigned to response patterns/health states considered worse than death. The best pattern is assigned the index value of 1.0; the worst pattern is assigned an index value of -0.594. Between-group differences in regression-predicted change from baseline score were estimated for the index. LS Mean value was controlled for Treatment, visit, Treatment*Visit and baseline.
Time Frame: From Randomization Date through End of Study (Up to 32 Months)
Population: All randomized participants who received at least one dose of study drug and with a baseline and at least 1 post-baseline result.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Abemaciclib | Erlotinib
Number analyzed (Participants) | 270 | 183
units on a scale | -0.08 (0.01) | -0.08 (0.02)
Statistical Analysis 1: Comparison: Abemaciclib vs Erlotinib; Test type: Superiority; p = 0.951, Mixed Models Analysis; Analyzed By Type 3 sums of squares, Change from Baseline = Treatment + Visit + Treatment*Visit + Baseline; LS Mean Change Difference = -0.00, 95% CI 2-sided [-0.05 to 0.05], Standard Error of Mean 0.02

7. Secondary Outcome: Resource Utilization: Percentage of Participants Who Are Hospitalized
Description: Resource utilization is the percentage of participants who was hospitalized.
Time Frame: From Randomization Date through End of Study (Up to 32 Months)
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Abemaciclib | Erlotinib
Number analyzed (Participants) | 265 | 175
percentage of participants | 40.4 | 22.9

ADVERSE EVENTS:
Time Frame: From Baseline to End of Study (Up to 47 Months)
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Abemaciclib | Erlotinib
All-Cause Mortality (participants affected / at risk) | 186/265 | 123/175
Serious Adverse Events (participants affected / at risk) | 112/265 | 43/175
Other Adverse Events (participants affected / at risk) | 247/265 | 161/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib (N=265) | Erlotinib (N=175)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 3 (3)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (7) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (6) | 2 (2)
Asthenia (General disorders) | 2 (4) | 0 (0)
Death (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 3 (3) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (3) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 3 (4) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 13 (15) | 6 (9)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia fungal (Infections and infestations) | 1 (2) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 2 (2)
Sepsis pasteurella (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 1 (2)
Skin infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chemical poisoning (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (6) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (2) | 0 (0)
Blood creatinine increased (Investigations) | 2 (6) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 3 (5) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 10 (12) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2) | 2 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 2 (2) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (3) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 2 (3) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 3 (4) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 10 (15) | 1 (1)
Anuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (11)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (3)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (4)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 1 (2)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib (N=265) | Erlotinib (N=175)
Anaemia (Blood and lymphatic system disorders) | 87 (163) | 23 (30)
Neutropenia (Blood and lymphatic system disorders) | 19 (44) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 17 (25) | 1 (3)
Abdominal pain (Gastrointestinal disorders) | 30 (34) | 8 (8)
Constipation (Gastrointestinal disorders) | 29 (32) | 15 (17)
Diarrhoea (Gastrointestinal disorders) | 169 (331) | 69 (100)
Nausea (Gastrointestinal disorders) | 94 (127) | 30 (33)
Stomatitis (Gastrointestinal disorders) | 14 (14) | 10 (10)
Vomiting (Gastrointestinal disorders) | 61 (89) | 15 (15)
Asthenia (General disorders) | 44 (82) | 13 (16)
Fatigue (General disorders) | 73 (132) | 29 (38)
Non-cardiac chest pain (General disorders) | 15 (17) | 7 (7)
Pyrexia (General disorders) | 33 (40) | 11 (11)
Aspartate aminotransferase increased (Investigations) | 15 (26) | 7 (8)
Blood creatinine increased (Investigations) | 45 (81) | 2 (2)
Neutrophil count decreased (Investigations) | 40 (130) | 2 (4)
Platelet count decreased (Investigations) | 42 (103) | 5 (7)
Weight decreased (Investigations) | 42 (54) | 16 (22)
White blood cell count decreased (Investigations) | 28 (83) | 4 (6)
Decreased appetite (Metabolism and nutrition disorders) | 95 (133) | 42 (52)
Dehydration (Metabolism and nutrition disorders) | 15 (18) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 18 (24) | 8 (15)
Hypokalaemia (Metabolism and nutrition disorders) | 22 (31) | 9 (10)
Hyponatraemia (Metabolism and nutrition disorders) | 17 (37) | 6 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (15) | 11 (15)
Dizziness (Nervous system disorders) | 18 (19) | 5 (6)
Headache (Nervous system disorders) | 24 (29) | 11 (12)
Insomnia (Psychiatric disorders) | 15 (16) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 38 (45) | 21 (22)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 53 (74) | 22 (26)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 16 (17) | 4 (4)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (4) | 46 (68)
Dry skin (Skin and subcutaneous tissue disorders) | 14 (14) | 26 (35)
Pruritus (Skin and subcutaneous tissue disorders) | 17 (22) | 18 (27)
Rash (Skin and subcutaneous tissue disorders) | 11 (14) | 42 (68)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (3):
  • Study Protocol: Protocol (2014-05-13): https://cdn.clinicaltrials.gov/large-docs/31/NCT02152631/Prot_001.pdf
  • Study Protocol: Protocol (e) (2016-12-20): https://cdn.clinicaltrials.gov/large-docs/31/NCT02152631/Prot_002.pdf
  • Statistical Analysis Plan (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/31/NCT02152631/SAP_000.pdf